CLINICAL TRIAL: NCT00056056
Title: A Randomized, Open-Label Phase III Trial to Evaluate the Efficacy and Safety of Bexarotene (Targretin) Capsules Combined With PUVA, Compared to PUVA Treatment Alone in Patients With Mycosis Fungoides
Brief Title: Ultraviolet Light Therapy Using Methoxsalen With or Without Bexarotene in Treating Patients With Mycosis Fungoides
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: poor accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-21011; 2004-003701-24 (EudraCT Number)
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Lymphoma
Keywords: stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome
MeSH Terms: conditions — Lymphoma; Mycosis Fungoides; Sezary Syndrome | interventions — Bexarotene; Methoxsalen; Ultraviolet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bexarotene and PUVA (Experimental)
  Interventions: Drug: bexarotene; Drug: methoxypsoralen; Procedure: UV light therapy
- PUVA (Active Comparator)
  Interventions: Drug: methoxypsoralen; Procedure: UV light therapy

INTERVENTIONS:
Drug: bexarotene — The recommended initial dosage of Bexarotene (75 mg Bexarotene capsules to be administered according to body surface area) for patients entered in this trial is 300 mg/m2 /once a day, taken orally, till CCR, PD, unacceptable toxicity, 16 weeks of treatment, whichever comes first
  Arms: Bexarotene and PUVA
Drug: methoxypsoralen — The dose of methoxypsoralen, as conventional capsules or liquid-filled capsules, is based on the patient's weight. The standard dose of 0.6 mg/kg will be given to all patients three times weekly - Increasing dose of PUVA according to a set protocol after a Minimal Phototoxic Dose (MPD) testing.
Procedure: UV light therapy — Initial UVA light exposure times should be based on the minimal phototoxic dose (MPD) for the specific light source being used. MPD can be determined by irradiating several skin areas 2 cm in diameter with varying light exposure times and determining the exposure time that produces erythema at 72 hours. The initial dose of UVA administered will be 70% of the MPD. The dose of UVA for the subsequent UVA sessions will be increased according to a standard protocol consisting of 20% increments with each successive treatment session depending on the presence of erythema.

SUMMARY:
RATIONALE: Ultraviolet light therapy uses light and drugs that make cancer cells more sensitive to light to kill tumor cells. It is not yet known whether ultraviolet light therapy is more effective with or without bexarotene in treating mycosis fungoides.

PURPOSE: Randomized phase III trial to compare the effectiveness of ultraviolet light therapy using methoxsalen with or without bexarotene in treating patients who have mycosis fungoides.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine if ultraviolet A light therapy with methoxsalen (PUVA) with or without bexarotene yields a significantly higher overall response rate in patients with mycosis fungoides.
* Compare the overall response rate (CCR and partial response) in patients treated with these regimens.
* Compare the duration of CCR and time to relapse of patients treated with these regimens.
* Compare the number of PUVA sessions necessary to achieve a CCR in these patients.
* Determine the percentage of dropouts by patients treated with these regimens.
* Determine the safety of these regimens in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to participating center, age (60 and under vs over 60), and stage of disease (IB vs IIA). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive PUVA comprising oral methoxsalen given 2 hours before whole body ultraviolet A therapy. PUVA is given 3 times per week.
* Arm II: Patients receive oral bexarotene once daily and PUVA as in arm I. In both arms, treatment repeats for up to 16 weeks in the absence of complete clinical response, disease progression, or unacceptable toxicity.

Patients are followed every 8 weeks until the first documented progression or relapse.

PROJECTED ACCRUAL: A total of 145 patients will be accrued for this study within 25 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed mycosis fungoides

  * Stage IB or IIA
  * Confirmed by current or prior diagnostic lesion biopsy

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* WBC at least 2,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN

Renal

* Creatinine no greater than 2 times ULN
* Calcium no greater than 11.5 mg/dL

Cardiovascular

* No New York Heart Association grade III or IV cardiac insufficiency

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study participation* NOTE: *Women using hormonal contraception must also use a non-hormonal treatment
* Fasting triglycerides normal (prior antilipemic agents allowed to reach normalization)
* Willing and able to avoid prolonged exposure to the sun

  * Willing to limit sun exposure on day of PUVA therapy
* No prior intolerance of or unresponsiveness to PUVA therapy
* No other prior or concurrent malignant tumor except adequately treated carcinoma in situ of the cervix or basal cell or squamous cell skin cancer
* No prior pancreatitis
* No other concurrent serious illness or infection that would preclude study participation
* No concurrent excessive alcohol consumption
* No photosensitivity due to intrinsic (e.g., lupus) or extrinsic (e.g., photosensitive drugs) factors
* No psychological, familial, sociological, or geographical condition that would preclude study compliance
* No known contraindications to study drug
* No known hypersensitivity to retinoids or hypervitaminosis A
* No uncontrolled diabetes mellitus
* No uncontrolled thyroid disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 months since prior interferon therapy

Chemotherapy

* No prior systemic combination chemotherapy
* No prior participation in another study of bexarotene
* At least 3 months since prior topical chemotherapy

Endocrine therapy

* At least 1 month since prior topical corticosteroids

Radiotherapy

* At least 6 months since prior total skin electron beam therapy
* At least 1 month since prior superficial radiotherapy

Surgery

* Not specified

Other

* At least 30 days since prior participation in another investigational drug study
* At least 3 months since prior photopheresis
* At least 1 month since prior UVB/PUVA phototherapy
* At least 1 month since prior retinoid class drugs
* At least 1 month since prior beta-carotene compounds
* At least 1 month since other prior topical medications (e.g., tar baths)
* No prior participation in this study
* No other concurrent anticancer therapy
* No other concurrent investigational drug therapy
* No concurrent drugs associated with pancreatic toxicity or known to increase triglyceride concentrations

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2003-01; Primary Completion 2010-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Overall response rate (complete clinical response [CCR) and partial response [PR]) | 35 months after first patient in

SECONDARY OUTCOMES:
Cumulative dose of UVA required to achieve CCR | 35 months after first patient in
Number of PUVA sessions necessary to achieve a CCR | 35 months after first patient in
Duration of CCR as measured by Logrank every 4 weeks during treatment and then every 8 weeks until progression | 35 months after first patient in
Time to relapse | 35 months after first patient in
Safety as assessed by CTC v2.0 every 4 weeks during treatment, then every 8 weeks | 35 months after first patient in
Percentage of dropouts as measured by the percentage of cases not completing treatment due to toxicity at the completion of treatment | 35 months after first patient in

CONTACTS AND LOCATIONS:
Overall Officials: Sean J. Whittaker, MD, Study Chair — St. Thomas' Hospital
Locations (28):
- Austria (2):
  - Karl-Franzens-University Graz, Graz
  - Allgemeines Krankenhaus - Universitatskliniken, Vienna
- Belgium (2):
  - Ghent University, Ghent
  - U.Z. Gasthuisberg, Leuven
- Bispebjerg Hospital, Copenhagen, Denmark
- Helsinki University Central Hospital, Helsinki, Finland
- France (2):
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - CHR Hotel Dieu, Nantes
- Germany (5):
  - Klinikum der Stadt Mannheim, Mannheim
  - Klinikum Minden, Minden
  - Hospital Universitario Insular de Gran Canaria, Tübingen
  - Southwest German Cancer Center at Eberhard-Karls-University, Tübingen
  - Medizinische Klinik und Poliklinik II - Universitaetsklinikum Wuerzburg, Würzburg
- Hungary (2):
  - Semmelweis University, Budapest
  - County Hospital, Kaposvár
- Rabin Medical Center - Beilinson Campus, Petah Tikva, Israel
- Italy (3):
  - Spedali Civili di Brescia, Brescia
  - Istituto Dermopatico Dell' Immacolata, Rome
  - Universita di Torino, Turin
- Leiden University Medical Center, Leiden, Netherlands
- Spain (5):
  - Hospital de la Santa Cruz i Sant Pau, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Nuestra Senora de la Candelaria, Santa Cruz de Tenerife
- UniversitaetsSpital Zuerich, Zurich, Switzerland
- United Kingdom (2):
  - St. Thomas' Hospital, London, England
  - Royal Infirmary of Edinburgh at Little France, Edinburgh, Scotland

REFERENCES:
- [Derived] Whittaker S, Ortiz P, Dummer R, Ranki A, Hasan B, Meulemans B, Gellrich S, Knobler R, Stadler R, Karrasch M. Efficacy and safety of bexarotene combined with psoralen-ultraviolet A (PUVA) compared with PUVA treatment alone in stage IB-IIA mycosis fungoides: final results from the EORTC Cutaneous Lymphoma Task Force phase III randomized clinical trial (NCT00056056). Br J Dermatol. 2012 Sep;167(3):678-87. doi: 10.1111/j.1365-2133.2012.11156.x. PMID 22924950